CLINICAL TRIAL: NCT00445224
Title: Comparison of Early Hip Strengthening to Early Quadriceps Strengthening in the Treatment of Females With Patellofemoral Pain
Brief Title: Comparing Rehabilitation Programs for Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Timothy Uhl (Other)
Responsible Party: Sponsor-Investigator, Timothy Uhl, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 07-0138-F2L
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Results first posted 2010-08-05 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Knee pain; Rehabilitation
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hip Progressive Resistive Exercises (Experimental): Exercises targeting hip musculature such as hip abduction and hip external rotation that was progressed by increased resistance following typical progressive resistive exercise approach.
  Interventions: Other: Hip Progressive Resistive Exercise
- Quad Progressive Resistive Exercises (Active Comparator): Exercises targeting quadriceps musculature such as quadriceps isometric setting, terminal knee extensions, and straight leg raises that was progressed by increased resistance following typical progressive resistive exercise approach..
  Interventions: Other: Quad Progressive Resistive Exercises

INTERVENTIONS:
Other: Hip Progressive Resistive Exercise — Hip Progressive Resistance Exercise program will be carried out by subjects under supervision once a week and then performed at home 2 additional times at home without supervision. Exercises focus on strengthening hip abduction ad external rotation musculature.
  Arms: Hip Progressive Resistive Exercises
Other: Quad Progressive Resistive Exercises — Quad Progressive Resistive Exercise program will be carried out by subjects under supervision once a week and then performed at home 2 additional times at home without supervision. Exercises focus on strengthening quadriceps musculature with straight leg raises and quadriceps isometrics.
  Arms: Quad Progressive Resistive Exercises

SUMMARY:
Patellofemoral pain syndrome (PFPS) is a common knee disorder affecting physically active people. Despite the growing base of support for the early introduction of hip strengthening exercises into the rehabilitation of PFPS, there have been few randomized clinical trials comparing isolated hip to isolated quadriceps strengthening. The purpose of this study is to determine how different exercises affect pain, strength, muscle activity, and function in female subjects with patellofemoral pain. The researchers hypothesize that females diagnosed with PFPS who initially participate in a hip strengthening program will report a greater perceived level of function, greater strength, less pain, and improved neuromuscular activity than those who participate in a progressive quadriceps strengthening intervention.

DETAILED DESCRIPTION:
Methods: Thirty-three females with PFPS will perform either initial hip strengthening (hip group) or initial quadriceps strengthening (quad group) for 4 weeks, prior to 4 weeks of a similar program of functional weight-bearing exercises. Self-reported pain, function, and functional strength were measured. Isometric strength was assessed for hip abductors, external rotators, and knee extensors. A mixed-model analysis of variance will be used to determine group differences over time.

ELIGIBILITY:
Inclusion Criteria:

* anterior or retropatellar knee pain reported during at least 2 of the following activities: ascending and descending stairs, hopping and running, squatting, kneeling, and prolonged sitting
* insidious onset of symptoms not related to trauma
* pain with compression of the patella
* pain on palpation of the patellar facets

Exclusion Criteria:

* symptoms present for less than one month
* clinical evidence of other knee pathology
* history of recent knee surgery within past one year
* history of patellar dislocations or subluxations
* current significant injury affecting other lower extremity joints

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Uhl, PhD, ATC, PT, Study Chair — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided
willing to share strength and patient reported outcome data at pre, mid, and post testing time points.

REFERENCES:
- [Derived] Dolak KL, Silkman C, Medina McKeon J, Hosey RG, Lattermann C, Uhl TL. Hip strengthening prior to functional exercises reduces pain sooner than quadriceps strengthening in females with patellofemoral pain syndrome: a randomized clinical trial. J Orthop Sports Phys Ther. 2011 Aug;41(8):560-70. doi: 10.2519/jospt.2011.3499. Epub 2011 Jun 7. PMID 21654093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 33 females with anterior knee pain (PFPS) volunteered to participate in this study. Enrollment began August 2007 and last subject was enrolled in August 2009.
Pre-assignment Details: Subjects were evaluated for PFPS using the following:(1)anterior knee pain reported during at least 2 activities: stair climbing, running, squatting, kneeling, and prolonged sitting;(2)insidious onset of symptoms ;(3)pain with compression of the patella; and(4)pain on palpation of patellar facets. Only three patients were excluded during study.
Groups:
- Hip Strengthening Then Combined Exercises: Performed hip strengthening exercises for 4 weeks prior to crossing over to a combined hip and quadricep rehabilitation program
- Quadricep Group Then Combined Exercises: Performed quadricep strengthening exercises for 4 weeks prior to crossing over to a combined hip and quadricep rehabilitation program
Period: Specific Exercises
Arm/Group | Hip Strengthening Then Combined Exercises | Quadricep Group Then Combined Exercises
Started | 17 | 16
Baseline | 17 | 16
4 Weeks | 14 (Participants withdrew due to time conflicts) | 13 (Participants withdrew due to time conflicts)
Completed | 13 (No adverse event occurred) | 13 (No adverse event occurred)
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Withdrawal by Subject | 1 | 0
Period: Combined Exercises
Arm/Group | Hip Strengthening Then Combined Exercises | Quadricep Group Then Combined Exercises
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hip Strengthening Then Combined Exercises | Quadricep Group Then Combined Exercises | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.6 (5.3) | 25.7 (5.9) | 25 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Pain Scale (Describing Worst Pain Felt During the Past Week)
Description: 0 to 10 cm line with 0 representing no pain and 10 representing severe pain
Time Frame: weekly
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Hip Strengthening Then Combined Exercises | Quadricep Group Then Combined Exercises
Number analyzed (Participants) | 17 | 16
centimeter | 4.5 (2.5) | 4.2 (2.2)

2. Primary Outcome: Subjective Function by Lower Extremity Functional Scale Report Form
Time Frame: Baseline, Mid-Intervention, and Post-Intervention
Reporting Status: Not Posted

3. Secondary Outcome: Strength by Isometric Dynamometer
Time Frame: Baseline, Mid, and Post-Intervention
Reporting Status: Not Posted

4. Secondary Outcome: Neuromuscular Activity by Surface Electromyographical Amplitude During Stair Descent
Time Frame: Baseline, Mid and Post-Intervention
Reporting Status: Not Posted

5. Secondary Outcome: Objective Function by Step-down Task for 30 Seconds
Time Frame: Baseline, Mid, and Post-Intervention
Reporting Status: Not Posted

6. Secondary Outcome: Hip Abduction Strength
Description: Side lying Hip Abduction maximal muscular contraction with a hand held dynamometer
Time Frame: 8 week
Measure: Mean (Standard Deviation); unit: (Newton*meters)/(Weight*Height)
Arm/Group | Hip Strengthening Then Combined Exercises | Quadricep Group Then Combined Exercises
Number analyzed (Participants) | 17 | 16
(Newton*meters)/(Weight*Height) | 6.6 (.9) | 6.2 (1.8)
Statistical Analysis 1: Comparison: Hip Strengthening Then Combined Exercises vs Quadricep Group Then Combined Exercises; Test type: Superiority or Other; p = .041, ANOVA

7. Primary Outcome: Visual Analog Pain Scale
Description: Visual analog pain scale at end of intervention. 0 to 10 cm line with 0 representing no pain and 10 representing severe pain
Time Frame: 8 week
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Hip Strengthening Then Combined Exercises | Quadricep Group Then Combined Exercises
Number analyzed (Participants) | 17 | 16
centimeters | 2.4 (2.8) | 2.6 (2.0)
Statistical Analysis 1: Comparison: Hip Strengthening Then Combined Exercises vs Quadricep Group Then Combined Exercises; Repeated measures ANOVA for group and time; Test type: Superiority or Other; p = .049, ANOVA

ADVERSE EVENTS:
Time Frame: During the study and for 6 months following the study
Arm/Group | Hip Strengthening Then Combined Exercises | Quadricep Group Then Combined Exercises
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed. Intention to treat analysis, last score carried forward, was used to analyze all outcome data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes